CLINICAL TRIAL: NCT04474392
Title: Sputum Studies of Anti-Citrullinated Protein Antibodies (ACPA) and Rheumatoid Arthritis (RA) Origins
Acronym: SPARO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20-0206; 1R01AR076450-01 (NIH)
Record Dates: First submitted 2020-06-29; First posted 2020-07-16 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, saliva, and sputum samples are collected for this study. The blood, saliva, and sputum samples are stored in -80 freezers at the Barbara Davis Center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- At-Risk (N=180): 1. No evidence of inflammatory arthritis on clinical examination AND
  2. At elevated risk for RA based on familial or serologic risk
     * Familial risk includes having a first degree relatives (FDRs) with RA
     * Serologic risk includes asymptomatic serum ACPA positivity
  There will be 1 study visit per year for 3 years; for a subset of 30 of these participants, there will be an additional 3 quarterly visits in one year.
  Study Procedures (Baseline & Follow-up):
  * Questionnaires
  * Physical and joint exam
  * Measurement of participants' height, weight
  * Blood and sputum collection
  Interventions: Other: N/A (Observational Study)
- Healthy Controls (N=120): 1. No history of RA
  2. No FDRs with RA
  3. No systemic use of immunosuppressants for autoimmune disease
  Participants will return for 1 follow-up visit, approximately 1 year after their baseline visit.
  Study Procedures (Baseline & Follow-up):
  * Questionnaires
  * Physical and joint exam
  * Measurement of participants' height, weight
  * Blood and sputum collection
  Interventions: Other: N/A (Observational Study)
- RA Diagnosis (N=40): 1. Classified RA by 1987 ACR and/or 2010 ACR/EULAR RA classification criteria (confirmed by medical chart review) OR
  2. Diagnosed with RA by a board-certified rheumatologist (confirmed by medical chart review)
  Participants will return for 1 follow-up visit, approximately 1 year after their baseline visit.
  Study Procedures (Baseline & Follow-up):
  * Questionnaires
  * Physical and joint exam
  * Measurement of participants' height, weight
  * Blood and sputum collection
  Interventions: Other: N/A (Observational Study)

INTERVENTIONS:
Other: N/A (Observational Study) — Observational study, no intervention will be administered.

SUMMARY:
The study is designed to learn more about the causes of rheumatoid arthritis (RA). People who get RA have elevated protein markers called autoantibodies in their blood years before initial symptoms of arthritis. The goal of this study is to learn more about how autoantibodies in RA might be related to inflammation in the lungs.

DETAILED DESCRIPTION:
The Specific Aims of This Study Are As Follows:

1. Identify whether sputum anti-CCP predicts incident RA
2. Determine the effect of inflammatory cytokines on the induction of NETosis in sputum neutrophils
3. Determine the role of sputum macrophage phagocytosis in NET clearance <br> The knowledge gained from this study will improve the overall understanding of the development of RA. It is anticipated that these findings will improve the field's understanding of how best to screen for RA risk and target RA prevention. This study could support future lung-targeted prevention strategies for RA that could avoid the administration of systemic toxic therapies. Such potential prevention interventions could be implemented in subjects at risk for RA in order to prevent the irreversible joint damage that can occur in the later stages of clinically-apparent RA.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 100 years;
* At-Risk for RA, RA diagnosed, and Healthy Control subjects will be included in the study until recruitment goals are met for each group.

At-Risk:

1. No evidence of inflammatory arthritis on clinical examination AND
2. At elevated risk for RA based on familial or serologic risk

   * Familial risk includes having a first degree relatives (FDRs) with RA
   * Serologic risk includes asymptomatic serum ACPA positivity

Healthy Controls :

1. No history of RA
2. No FDRs with RA
3. No systemic use of immunosuppressants for autoimmune disease

RA Diagnosis:

1. Classified RA by 1987 ACR and/or 2010 ACR/EULAR RA classification criteria (confirmed by medical chart review) OR
2. Diagnosed with RA by a board-certified rheumatologist (confirmed by medical chart review)

Exclusion Criteria:

1. Currently pregnant or planning to become pregnant during the sample collection period of the study
2. Exacerbation of underlying obstructive lung disease within the past 1 month
3. Known FEV1 <1 liter
4. Oxygen requirement >2 liters at rest
5. Participants with health acuity or behavioral health concerns leaving them unable to participate in the current research

Note: If a subject temporarily does not meet inclusion criteria but is interested in participating, he/she may participate once inclusion criteria have been met.

If interested, please take a few minutes to complete the screening questionnaire for this study opportunity. You may open the survey in your web browser by clicking the link below:

https://is.gd/SPAROscreen

If the link above does not work, try copying the link below into your web browser:

https://redcap.ucdenver.edu/surveys/?s=3WM8WH3WKK

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit subjects from 1) the Denver site of the SERA project (COMIRB #01-0675); 2) local rheumatology clinics, including the University of Colorado Hospital (UCH), Denver Health, National Jewish Health (NJH), and the Denver Arthritis Clinic; 3) local health clinics at UCH; and 4) local advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-07-14 (Estimated); Study Completion 2025-07-14 (Estimated)

PRIMARY OUTCOMES:
Sputum anti-CCP antibodies predicting incident RA | 1-3 years per participant (depending on group); study visits x1 per year, with option for 3 additional visits over 1 year for a subgroup of participants.
  *Sputum anti-CCP antibodies every year for 3 years (subjects At-Risk for RA); to identify whether sputum anti-CCP predicts incident RA

SECONDARY OUTCOMES:
Effect of inflammatory cytokines on the induction of NETosis in sputum neutrophils | 1-3 yrs / participant; At-Risk Group: Baseline Visit & 2 Follow-up Annual Visits (w/ potential to have 3 additional visits in 1 year); Healthy Controls & RA Diagnosed: Baseline Visit & 1 Follow-up Visit, approximately 1 year later
  *Determine the effect of inflammatory cytokines on the induction of NETosis in sputum neutrophils
The role of sputum macrophage phagocytosis in NET clearance | 1-3 years / participant; At-Risk Group: Baseline Visit & 2 Follow-up Annual Visits (w/ potential to have 3 additional visits in 1 year); Healthy Controls & RA Diagnosed: Baseline Visit & 1 Follow-up Visit, approximately 1 year later
  *Determine the role of sputum macrophage phagocytosis in NET clearance among At-Risk, healthy, & RA subjects

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Demoruelle, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver (Anschutz Medical Campus), Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Allaire S, Wolfe F, Niu J, Lavalley MP. Contemporary prevalence and incidence of work disability associated with rheumatoid arthritis in the US. Arthritis Rheum. 2008 Apr 15;59(4):474-80. doi: 10.1002/art.23538. PMID 18383413
- [Background] van der Woude D, Young A, Jayakumar K, Mertens BJ, Toes RE, van der Heijde D, Huizinga TW, van der Helm-van Mil AH. Prevalence of and predictive factors for sustained disease-modifying antirheumatic drug-free remission in rheumatoid arthritis: results from two large early arthritis cohorts. Arthritis Rheum. 2009 Aug;60(8):2262-71. doi: 10.1002/art.24661. PMID 19644846
- [Background] Ogdie A, Haynes K, Troxel AB, Love TJ, Hennessy S, Choi H, Gelfand JM. Risk of mortality in patients with psoriatic arthritis, rheumatoid arthritis and psoriasis: a longitudinal cohort study. Ann Rheum Dis. 2014 Jan;73(1):149-53. doi: 10.1136/annrheumdis-2012-202424. Epub 2012 Dec 21. PMID 23264338
- [Background] Birnbaum H, Pike C, Kaufman R, Marynchenko M, Kidolezi Y, Cifaldi M. Societal cost of rheumatoid arthritis patients in the US. Curr Med Res Opin. 2010 Jan;26(1):77-90. doi: 10.1185/03007990903422307. PMID 19908947
- [Background] Deane KD, Striebich CC, Holers VM. Editorial: Prevention of Rheumatoid Arthritis: Now Is the Time, but How to Proceed? Arthritis Rheumatol. 2017 May;69(5):873-877. doi: 10.1002/art.40061. Epub 2017 Apr 11. No abstract available. PMID 28217918
- [Background] Hunt L, Hensor EM, Nam J, Burska AN, Parmar R, Emery P, Ponchel F. T cell subsets: an immunological biomarker to predict progression to clinical arthritis in ACPA-positive individuals. Ann Rheum Dis. 2016 Oct;75(10):1884-9. doi: 10.1136/annrheumdis-2015-207991. Epub 2015 Dec 1. PMID 27613874
- [Background] Harre U, Georgess D, Bang H, Bozec A, Axmann R, Ossipova E, Jakobsson PJ, Baum W, Nimmerjahn F, Szarka E, Sarmay G, Krumbholz G, Neumann E, Toes R, Scherer HU, Catrina AI, Klareskog L, Jurdic P, Schett G. Induction of osteoclastogenesis and bone loss by human autoantibodies against citrullinated vimentin. J Clin Invest. 2012 May;122(5):1791-802. doi: 10.1172/JCI60975. Epub 2012 Apr 16. PMID 22505457
- [Background] Kuhn KA, Kulik L, Tomooka B, Braschler KJ, Arend WP, Robinson WH, Holers VM. Antibodies against citrullinated proteins enhance tissue injury in experimental autoimmune arthritis. J Clin Invest. 2006 Apr;116(4):961-73. doi: 10.1172/JCI25422. PMID 16585962
- [Background] Clavel C, Nogueira L, Laurent L, Iobagiu C, Vincent C, Sebbag M, Serre G. Induction of macrophage secretion of tumor necrosis factor alpha through Fcgamma receptor IIa engagement by rheumatoid arthritis-specific autoantibodies to citrullinated proteins complexed with fibrinogen. Arthritis Rheum. 2008 Mar;58(3):678-88. doi: 10.1002/art.23284. PMID 18311806
- [Background] Titcombe PJ, Wigerblad G, Sippl N, Zhang N, Shmagel AK, Sahlstrom P, Zhang Y, Barsness LO, Ghodke-Puranik Y, Baharpoor A, Hansson M, Israelsson L, Skriner K, Niewold TB, Klareskog L, Svensson CI, Amara K, Malmstrom V, Mueller DL. Pathogenic Citrulline-Multispecific B Cell Receptor Clades in Rheumatoid Arthritis. Arthritis Rheumatol. 2018 Dec;70(12):1933-1945. doi: 10.1002/art.40590. Epub 2018 Oct 18. PMID 29927106
- [Background] Engdahl C, Bang H, Dietel K, Lang SC, Harre U, Schett G. Periarticular Bone Loss in Arthritis Is Induced by Autoantibodies Against Citrullinated Vimentin. J Bone Miner Res. 2017 Aug;32(8):1681-1691. doi: 10.1002/jbmr.3158. Epub 2017 May 26. PMID 28425620
- [Background] Krishnamurthy A, Joshua V, Haj Hensvold A, Jin T, Sun M, Vivar N, Ytterberg AJ, Engstrom M, Fernandes-Cerqueira C, Amara K, Magnusson M, Wigerblad G, Kato J, Jimenez-Andrade JM, Tyson K, Rapecki S, Lundberg K, Catrina SB, Jakobsson PJ, Svensson C, Malmstrom V, Klareskog L, Wahamaa H, Catrina AI. Identification of a novel chemokine-dependent molecular mechanism underlying rheumatoid arthritis-associated autoantibody-mediated bone loss. Ann Rheum Dis. 2016 Apr;75(4):721-9. doi: 10.1136/annrheumdis-2015-208093. Epub 2015 Nov 26. PMID 26612338
- [Background] Wigerblad G, Bas DB, Fernades-Cerqueira C, Krishnamurthy A, Nandakumar KS, Rogoz K, Kato J, Sandor K, Su J, Jimenez-Andrade JM, Finn A, Bersellini Farinotti A, Amara K, Lundberg K, Holmdahl R, Jakobsson PJ, Malmstrom V, Catrina AI, Klareskog L, Svensson CI. Autoantibodies to citrullinated proteins induce joint pain independent of inflammation via a chemokine-dependent mechanism. Ann Rheum Dis. 2016 Apr;75(4):730-8. doi: 10.1136/annrheumdis-2015-208094. Epub 2015 Nov 27. PMID 26613766
- [Background] Demoruelle MK, Parish MC, Derber LA, Kolfenbach JR, Hughes-Austin JM, Weisman MH, Gilliland W, Edison JD, Buckner JH, Mikuls TR, O'Dell JR, Keating RM, Gregersen PK, Norris JM, Holers VM, Deane KD. Performance of anti-cyclic citrullinated Peptide assays differs in subjects at increased risk of rheumatoid arthritis and subjects with established disease. Arthritis Rheum. 2013 Sep;65(9):2243-52. doi: 10.1002/art.38017. PMID 23686569
- [Background] Rantapaa-Dahlqvist S, de Jong BA, Berglin E, Hallmans G, Wadell G, Stenlund H, Sundin U, van Venrooij WJ. Antibodies against cyclic citrullinated peptide and IgA rheumatoid factor predict the development of rheumatoid arthritis. Arthritis Rheum. 2003 Oct;48(10):2741-9. doi: 10.1002/art.11223. PMID 14558078
- [Background] Nielen MM, van Schaardenburg D, Reesink HW, van de Stadt RJ, van der Horst-Bruinsma IE, de Koning MH, Habibuw MR, Vandenbroucke JP, Dijkmans BA. Specific autoantibodies precede the symptoms of rheumatoid arthritis: a study of serial measurements in blood donors. Arthritis Rheum. 2004 Feb;50(2):380-6. doi: 10.1002/art.20018. PMID 14872479
- [Background] Brink M, Hansson M, Mathsson L, Jakobsson PJ, Holmdahl R, Hallmans G, Stenlund H, Ronnelid J, Klareskog L, Rantapaa-Dahlqvist S. Multiplex analyses of antibodies against citrullinated peptides in individuals prior to development of rheumatoid arthritis. Arthritis Rheum. 2013 Apr;65(4):899-910. doi: 10.1002/art.37835. PMID 23310951
- [Background] Ramos-Remus C, Castillo-Ortiz JD, Aguilar-Lozano L, Padilla-Ibarra J, Sandoval-Castro C, Vargas-Serafin CO, de la Mora-Molina H, Ramos-Gomez A, Sanchez-Ortiz A, Avila-Armengol H, Aceves-Avila FJ. Autoantibodies in prediction of the development of rheumatoid arthritis among healthy relatives of patients with the disease. Arthritis Rheumatol. 2015 Nov;67(11):2837-44. doi: 10.1002/art.39297. PMID 26245885
- [Background] Ford JA, Liu X, Marshall AA, Zaccardelli A, Prado MG, Wiyarand C, Lu B, Karlson EW, Schur PH, Deane KD, Sparks JA. Impact of Cyclic Citrullinated Peptide Antibody Level on Progression to Rheumatoid Arthritis in Clinically Tested Cyclic Citrullinated Peptide Antibody-Positive Patients Without Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2019 Dec;71(12):1583-1592. doi: 10.1002/acr.23820. PMID 30570827
- [Background] van de Stadt LA, Witte BI, Bos WH, van Schaardenburg D. A prediction rule for the development of arthritis in seropositive arthralgia patients. Ann Rheum Dis. 2013 Dec;72(12):1920-6. doi: 10.1136/annrheumdis-2012-202127. Epub 2012 Nov 23. PMID 23178208
- [Background] Kokkonen H, Mullazehi M, Berglin E, Hallmans G, Wadell G, Ronnelid J, Rantapaa-Dahlqvist S. Antibodies of IgG, IgA and IgM isotypes against cyclic citrullinated peptide precede the development of rheumatoid arthritis. Arthritis Res Ther. 2011 Feb 3;13(1):R13. doi: 10.1186/ar3237. PMID 21291540
- [Background] Rakieh C, Nam JL, Hunt L, Hensor EM, Das S, Bissell LA, Villeneuve E, McGonagle D, Hodgson R, Grainger A, Wakefield RJ, Conaghan PG, Emery P. Predicting the development of clinical arthritis in anti-CCP positive individuals with non-specific musculoskeletal symptoms: a prospective observational cohort study. Ann Rheum Dis. 2015 Sep;74(9):1659-66. doi: 10.1136/annrheumdis-2014-205227. Epub 2014 Apr 12. PMID 24728331
- [Background] van de Sande MG, de Hair MJ, van der Leij C, Klarenbeek PL, Bos WH, Smith MD, Maas M, de Vries N, van Schaardenburg D, Dijkmans BA, Gerlag DM, Tak PP. Different stages of rheumatoid arthritis: features of the synovium in the preclinical phase. Ann Rheum Dis. 2011 May;70(5):772-7. doi: 10.1136/ard.2010.139527. Epub 2010 Dec 21. PMID 21177292
- [Background] Demoruelle MK, Weisman MH, Simonian PL, Lynch DA, Sachs PB, Pedraza IF, Harrington AR, Kolfenbach JR, Striebich CC, Pham QN, Strickland CD, Petersen BD, Parish MC, Derber LA, Norris JM, Holers VM, Deane KD. Brief report: airways abnormalities and rheumatoid arthritis-related autoantibodies in subjects without arthritis: early injury or initiating site of autoimmunity? Arthritis Rheum. 2012 Jun;64(6):1756-61. doi: 10.1002/art.34344. Epub 2011 Dec 19. PMID 22183986
- [Background] Willis VC, Demoruelle MK, Derber LA, Chartier-Logan CJ, Parish MC, Pedraza IF, Weisman MH, Norris JM, Holers VM, Deane KD. Sputum autoantibodies in patients with established rheumatoid arthritis and subjects at risk of future clinically apparent disease. Arthritis Rheum. 2013 Oct;65(10):2545-54. doi: 10.1002/art.38066. PMID 23817979
- [Background] Demoruelle MK, Harrall KK, Ho L, Purmalek MM, Seto NL, Rothfuss HM, Weisman MH, Solomon JJ, Fischer A, Okamoto Y, Kelmenson LB, Parish MC, Feser M, Fleischer C, Anderson C, Mahler M, Norris JM, Kaplan MJ, Cherrington BD, Holers VM, Deane KD. Anti-Citrullinated Protein Antibodies Are Associated With Neutrophil Extracellular Traps in the Sputum in Relatives of Rheumatoid Arthritis Patients. Arthritis Rheumatol. 2017 Jun;69(6):1165-1175. doi: 10.1002/art.40066. Epub 2017 May 2. PMID 28182854
- [Background] Demoruelle MK, Bowers E, Lahey LJ, Sokolove J, Purmalek M, Seto NL, Weisman MH, Norris JM, Kaplan MJ, Holers VM, Robinson WH, Deane KD. Antibody Responses to Citrullinated and Noncitrullinated Antigens in the Sputum of Subjects With Rheumatoid Arthritis and Subjects at Risk for Development of Rheumatoid Arthritis. Arthritis Rheumatol. 2018 Apr;70(4):516-527. doi: 10.1002/art.40401. Epub 2018 Mar 2. PMID 29266801
- [Background] Fischer A, Solomon JJ, du Bois RM, Deane KD, Olson AL, Fernandez-Perez ER, Huie TJ, Stevens AD, Gill MB, Rabinovitch AM, Lynch DA, Burns DA, Pineiro IS, Groshong SD, Duarte Achcar RD, Brown KK, Martin RJ, Swigris JJ. Lung disease with anti-CCP antibodies but not rheumatoid arthritis or connective tissue disease. Respir Med. 2012 Jul;106(7):1040-7. doi: 10.1016/j.rmed.2012.03.006. Epub 2012 Apr 12. PMID 22503074
- [Background] Klareskog L, Stolt P, Lundberg K, Kallberg H, Bengtsson C, Grunewald J, Ronnelid J, Harris HE, Ulfgren AK, Rantapaa-Dahlqvist S, Eklund A, Padyukov L, Alfredsson L. A new model for an etiology of rheumatoid arthritis: smoking may trigger HLA-DR (shared epitope)-restricted immune reactions to autoantigens modified by citrullination. Arthritis Rheum. 2006 Jan;54(1):38-46. doi: 10.1002/art.21575. PMID 16385494
- [Background] Reynisdottir G, Karimi R, Joshua V, Olsen H, Hensvold AH, Harju A, Engstrom M, Grunewald J, Nyren S, Eklund A, Klareskog L, Skold CM, Catrina AI. Structural changes and antibody enrichment in the lungs are early features of anti-citrullinated protein antibody-positive rheumatoid arthritis. Arthritis Rheumatol. 2014 Jan;66(1):31-9. doi: 10.1002/art.38201. PMID 24449573
- [Background] Makrygiannakis D, Hermansson M, Ulfgren AK, Nicholas AP, Zendman AJ, Eklund A, Grunewald J, Skold CM, Klareskog L, Catrina AI. Smoking increases peptidylarginine deiminase 2 enzyme expression in human lungs and increases citrullination in BAL cells. Ann Rheum Dis. 2008 Oct;67(10):1488-92. doi: 10.1136/ard.2007.075192. Epub 2008 Apr 15. PMID 18413445
- [Background] Rangel-Moreno J, Hartson L, Navarro C, Gaxiola M, Selman M, Randall TD. Inducible bronchus-associated lymphoid tissue (iBALT) in patients with pulmonary complications of rheumatoid arthritis. J Clin Invest. 2006 Dec;116(12):3183-94. doi: 10.1172/JCI28756. PMID 17143328
- [Background] Quirke AM, Perry E, Cartwright A, Kelly C, De Soyza A, Eggleton P, Hutchinson D, Venables PJ. Bronchiectasis is a Model for Chronic Bacterial Infection Inducing Autoimmunity in Rheumatoid Arthritis. Arthritis Rheumatol. 2015 Sep;67(9):2335-42. doi: 10.1002/art.39226. PMID 26017630
- [Background] Janssen KM, de Smit MJ, Brouwer E, de Kok FA, Kraan J, Altenburg J, Verheul MK, Trouw LA, van Winkelhoff AJ, Vissink A, Westra J. Rheumatoid arthritis-associated autoantibodies in non-rheumatoid arthritis patients with mucosal inflammation: a case-control study. Arthritis Res Ther. 2015 Jul 9;17(1):174. doi: 10.1186/s13075-015-0690-6. PMID 26155788
- [Background] Reynisdottir G, Olsen H, Joshua V, Engstrom M, Forsslund H, Karimi R, Skold CM, Nyren S, Eklund A, Grunewald J, Catrina AI. Signs of immune activation and local inflammation are present in the bronchial tissue of patients with untreated early rheumatoid arthritis. Ann Rheum Dis. 2016 Sep;75(9):1722-7. doi: 10.1136/annrheumdis-2015-208216. Epub 2015 Nov 3. PMID 26530319
- [Background] Kinslow JD, Blum LK, Deane KD, Demoruelle MK, Okamoto Y, Parish MC, Kongpachith S, Lahey LJ, Norris JM, Robinson WH, Holers VM. Elevated IgA Plasmablast Levels in Subjects at Risk of Developing Rheumatoid Arthritis. Arthritis Rheumatol. 2016 Oct;68(10):2372-83. doi: 10.1002/art.39771. PMID 27273876
- [Background] Barra L, Bykerk V, Pope JE, Haraoui BP, Hitchon CA, Thorne JC, Keystone EC, Boire G; Catch Investigators. Anticitrullinated protein antibodies and rheumatoid factor fluctuate in early inflammatory arthritis and do not predict clinical outcomes. J Rheumatol. 2013 Aug;40(8):1259-67. doi: 10.3899/jrheum.120736. Epub 2013 Feb 1. PMID 23378461
- [Background] Brinkmann V, Reichard U, Goosmann C, Fauler B, Uhlemann Y, Weiss DS, Weinrauch Y, Zychlinsky A. Neutrophil extracellular traps kill bacteria. Science. 2004 Mar 5;303(5663):1532-5. doi: 10.1126/science.1092385. PMID 15001782
- [Background] Saffarzadeh M, Juenemann C, Queisser MA, Lochnit G, Barreto G, Galuska SP, Lohmeyer J, Preissner KT. Neutrophil extracellular traps directly induce epithelial and endothelial cell death: a predominant role of histones. PLoS One. 2012;7(2):e32366. doi: 10.1371/journal.pone.0032366. Epub 2012 Feb 28. PMID 22389696
- [Background] Khandpur R, Carmona-Rivera C, Vivekanandan-Giri A, Gizinski A, Yalavarthi S, Knight JS, Friday S, Li S, Patel RM, Subramanian V, Thompson P, Chen P, Fox DA, Pennathur S, Kaplan MJ. NETs are a source of citrullinated autoantigens and stimulate inflammatory responses in rheumatoid arthritis. Sci Transl Med. 2013 Mar 27;5(178):178ra40. doi: 10.1126/scitranslmed.3005580. PMID 23536012
- [Background] Sur Chowdhury C, Giaglis S, Walker UA, Buser A, Hahn S, Hasler P. Enhanced neutrophil extracellular trap generation in rheumatoid arthritis: analysis of underlying signal transduction pathways and potential diagnostic utility. Arthritis Res Ther. 2014 Jun 13;16(3):R122. doi: 10.1186/ar4579. PMID 24928093
- [Background] Pratesi F, Dioni I, Tommasi C, Alcaro MC, Paolini I, Barbetti F, Boscaro F, Panza F, Puxeddu I, Rovero P, Migliorini P. Antibodies from patients with rheumatoid arthritis target citrullinated histone 4 contained in neutrophils extracellular traps. Ann Rheum Dis. 2014 Jul;73(7):1414-22. doi: 10.1136/annrheumdis-2012-202765. Epub 2013 Jun 1. PMID 23727635
- [Background] Corsiero E, Bombardieri M, Carlotti E, Pratesi F, Robinson W, Migliorini P, Pitzalis C. Single cell cloning and recombinant monoclonal antibodies generation from RA synovial B cells reveal frequent targeting of citrullinated histones of NETs. Ann Rheum Dis. 2016 Oct;75(10):1866-75. doi: 10.1136/annrheumdis-2015-208356. Epub 2015 Dec 9. PMID 26659717
- [Background] Lloyd KA, Wigerblad G, Sahlstrom P, Garimella MG, Chemin K, Steen J, Titcombe PJ, Marklein B, Zhou D, Stalesen R, Ossipova E, Lundqvist C, Ekwall O, Ronnelid J, Mueller DL, Karlsson MCI, Kaplan MJ, Skriner K, Klareskog L, Wermeling F, Malmstrom V, Gronwall C. Differential ACPA Binding to Nuclear Antigens Reveals a PAD-Independent Pathway and a Distinct Subset of Acetylation Cross-Reactive Autoantibodies in Rheumatoid Arthritis. Front Immunol. 2019 Jan 4;9:3033. doi: 10.3389/fimmu.2018.03033. eCollection 2018. PMID 30662440
- [Background] Carmona-Rivera C, Carlucci PM, Moore E, Lingampalli N, Uchtenhagen H, James E, Liu Y, Bicker KL, Wahamaa H, Hoffmann V, Catrina AI, Thompson P, Buckner JH, Robinson WH, Fox DA, Kaplan MJ. Synovial fibroblast-neutrophil interactions promote pathogenic adaptive immunity in rheumatoid arthritis. Sci Immunol. 2017 Apr;2(10):eaag3358. doi: 10.1126/sciimmunol.aag3358. Epub 2017 Apr 14. PMID 28649674
- [Background] Skopelja-Gardner S, Jones JD, Rigby WFC. "NETtling" the host: Breaking of tolerance in chronic inflammation and chronic infection. J Autoimmun. 2018 Mar;88:1-10. doi: 10.1016/j.jaut.2017.10.008. PMID 29100671
- [Background] Dicker AJ, Crichton ML, Pumphrey EG, Cassidy AJ, Suarez-Cuartin G, Sibila O, Furrie E, Fong CJ, Ibrahim W, Brady G, Einarsson GG, Elborn JS, Schembri S, Marshall SE, Palmer CNA, Chalmers JD. Neutrophil extracellular traps are associated with disease severity and microbiota diversity in patients with chronic obstructive pulmonary disease. J Allergy Clin Immunol. 2018 Jan;141(1):117-127. doi: 10.1016/j.jaci.2017.04.022. Epub 2017 May 13. PMID 28506850
- [Background] Wright TK, Gibson PG, Simpson JL, McDonald VM, Wood LG, Baines KJ. Neutrophil extracellular traps are associated with inflammation in chronic airway disease. Respirology. 2016 Apr;21(3):467-75. doi: 10.1111/resp.12730. Epub 2016 Jan 25. PMID 26804470
- [Background] Grabcanovic-Musija F, Obermayer A, Stoiber W, Krautgartner WD, Steinbacher P, Winterberg N, Bathke AC, Klappacher M, Studnicka M. Neutrophil extracellular trap (NET) formation characterises stable and exacerbated COPD and correlates with airflow limitation. Respir Res. 2015 May 22;16(1):59. doi: 10.1186/s12931-015-0221-7. PMID 25994149
- [Background] Dworski R, Simon HU, Hoskins A, Yousefi S. Eosinophil and neutrophil extracellular DNA traps in human allergic asthmatic airways. J Allergy Clin Immunol. 2011 May;127(5):1260-6. doi: 10.1016/j.jaci.2010.12.1103. Epub 2011 Feb 18. PMID 21315435
- [Background] Lee J, Luria A, Rhodes C, Raghu H, Lingampalli N, Sharpe O, Rada B, Sohn DH, Robinson WH, Sokolove J. Nicotine drives neutrophil extracellular traps formation and accelerates collagen-induced arthritis. Rheumatology (Oxford). 2017 Apr 1;56(4):644-653. doi: 10.1093/rheumatology/kew449. PMID 28013195
- [Background] Porto BN, Stein RT. Neutrophil Extracellular Traps in Pulmonary Diseases: Too Much of a Good Thing? Front Immunol. 2016 Aug 15;7:311. doi: 10.3389/fimmu.2016.00311. eCollection 2016. PMID 27574522
- [Background] Frisell T, Holmqvist M, Kallberg H, Klareskog L, Alfredsson L, Askling J. Familial risks and heritability of rheumatoid arthritis: role of rheumatoid factor/anti-citrullinated protein antibody status, number and type of affected relatives, sex, and age. Arthritis Rheum. 2013 Nov;65(11):2773-82. doi: 10.1002/art.38097. PMID 23897126
- [Background] Hemminki K, Li X, Sundquist J, Sundquist K. Familial associations of rheumatoid arthritis with autoimmune diseases and related conditions. Arthritis Rheum. 2009 Mar;60(3):661-8. doi: 10.1002/art.24328. PMID 19248111
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Background] Arnett FC, Edworthy SM, Bloch DA, McShane DJ, Fries JF, Cooper NS, Healey LA, Kaplan SR, Liang MH, Luthra HS, et al. The American Rheumatism Association 1987 revised criteria for the classification of rheumatoid arthritis. Arthritis Rheum. 1988 Mar;31(3):315-24. doi: 10.1002/art.1780310302. PMID 3358796
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Snir O, Widhe M, Hermansson M, von Spee C, Lindberg J, Hensen S, Lundberg K, Engstrom A, Venables PJ, Toes RE, Holmdahl R, Klareskog L, Malmstrom V. Antibodies to several citrullinated antigens are enriched in the joints of rheumatoid arthritis patients. Arthritis Rheum. 2010 Jan;62(1):44-52. doi: 10.1002/art.25036. PMID 20039432
- [Background] Lood C, Blanco LP, Purmalek MM, Carmona-Rivera C, De Ravin SS, Smith CK, Malech HL, Ledbetter JA, Elkon KB, Kaplan MJ. Neutrophil extracellular traps enriched in oxidized mitochondrial DNA are interferogenic and contribute to lupus-like disease. Nat Med. 2016 Feb;22(2):146-53. doi: 10.1038/nm.4027. Epub 2016 Jan 18. PMID 26779811
- [Background] Gardner W, Mulvey EP, Shaw EC. Regression analyses of counts and rates: Poisson, overdispersed Poisson, and negative binomial models. Psychol Bull. 1995 Nov;118(3):392-404. doi: 10.1037/0033-2909.118.3.392. PMID 7501743
- [Background] Malickova K, Duricova D, Bortlik M, Hruskova Z, Svobodova B, Machkova N, Komarek V, Fucikova T, Janatkova I, Zima T, Lukas M. Impaired deoxyribonuclease I activity in patients with inflammatory bowel diseases. Autoimmune Dis. 2011;2011:945861. doi: 10.4061/2011/945861. Epub 2011 May 29. PMID 21687600